CLINICAL TRIAL: NCT03765541
Title: Dexamethasone Plus Salvage Chemotherapy Versus Salvage Chemotherapy Alone in Patients With First Relapsed or Refractory Acute Myeloid Leukemia: a Randomized, Controlled, Open-label, Multicenter, Phase III Study
Brief Title: Dexamethasone in Refractory or First Relapsed Acute Myeloid Leukemia
Acronym: DEXAML-03
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Despite a recruitment target that was not met, we managed to achieve more than 50% of inclusions and 33% of deaths, enabling us to carry out an initial analysis of the primary endpoint
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/17/0450
Record Dates: First submitted 2018-11-19; First posted 2018-12-05 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia
Keywords: dexamethasone; acute myeloid leukemia; relapse; refractory; azacitidine; amsacrine; cytarabine; randomized controlled trial
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute | interventions — Dexamethasone; Amsacrine; Cytarabine; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard salvage therapy + dexamethasone (Experimental): Intensive chemotherapy amsacrine-cytarabine or azacitidine according to the investigator's willingness in combination with dexamethasone
  Interventions: Drug: Dexamethasone; Drug: Amsacrine; Drug: Cytarabine; Drug: Azacitidine
- Standard salvage therapy alone (Active Comparator): Intensive chemotherapy amsacrine-cytarabine or azacitidine according to the investigator's willingness
  Interventions: Drug: Amsacrine; Drug: Cytarabine; Drug: Azacitidine

INTERVENTIONS:
Drug: Dexamethasone — In combination with intensive chemotherapy amsacrine-cytarabine:
  * Induction (1 cycle): 10 mg/12h from Day 1 to Day 3 of cycle (2 infusions/24h, slow IV [10 minutes])
  * Consolidation (3 cycles): 10 mg/12h from Day 1 to Day 3 of each cycle (2 infusions/24h, slow IV [10 minutes])
  In combination with azacitidine:
  * Cycle 1: 20 mg/24h from Day 1 to Day 3 of cycle (1 infusion/24h, slow IV [10 minutes]).
  * Subsequent cycles: 20 mg/24h on Day 1 of each cycle (1 infusion/24h, slow IV [10minutes]).
  Arms: Standard salvage therapy + dexamethasone
Drug: Amsacrine — * Induction (1 cycle): 200 mg/m2/24h from Day 1 to Day 3 of cycle (slow IV [3 hours])
  * Consolidation (3 cycles): 200 mg/m2/24h on Day 1 of each cycle (slow IV [3 hours])
Drug: Cytarabine — Patients < 60 years of age:
  * Induction (1 cycle): 3 g/m2/12h from Day 1 to Day 4 of cycle (2 infusions/24h, slow IV [2 hours])
  * Consolidation (3 cycles): 3 g/m2/12h from Day 1 to Day 3 of each cycle (2 infusions/24h, slow IV [2 hours]) Note: If the investigators believe that there is an undue risk for the safety of a patient under 60 years of age with comorbidity in receiving a dose level of 3 g/m2/12h, the dose may be reduced to 1 g/m2/12h
Drug: Azacitidine — 75 mg/m2/24h from Day 1 to Day 7 of each cycle [or from Day 1 to Day 5 and from Day 8 to Day 9 of each cycle] (SC)

SUMMARY:
Recent preclinical and retrospective clinical data have suggested that dexamethasone might sensitize leukemic cells to chemotherapy-induced cell death and thus limit the risk of leukemic regrowth and relapse. Moreover, it has been experimentally shown that leukemic cells in acute myeloid leukemia patients who relapse become sensitive to glucocorticoids treatment highlighting a novel potential role for dexamethasone in relapsed or refractory acute myeloid leukemia (R/R).

This study was designed to determine whether adding dexamethasone to standard salvage therapy in the treatment of relapsed/refractory acute myeloid leukemia in adult patients (intensive chemotherapy amsacrine-cytarabine or azacitidine according to investigator's willingness) results in a significant improvement of the overall survival.

DETAILED DESCRIPTION:
The prognosis for patients with relapsed or refractory acute myeloid leukemia is poor ; median survival is less than 1 year. High-dose cytarabine monotherapy or cytarabine-based combination regimens are often used as salvage therapy with limited efficacy. A recent retrospective study has shown that the addition of dexamethasone to intensive chemotherapy was significantly associated with better disease-free and overall survival in hyperleukocytic acute myeloid leukemia patients. The gene signatures of some molecular subgroups of acute myeloid leukemia were highly enriched in genes responsive to dexamethasone, including acute myeloid leukemia with NPM1 mutations which were particularly sensitive to the antileukemic activity of dexamethasone both in vitro and in vivo. Moreover, three recent preclinical studies have shown that cytarabine-resistant or RUNX1-mutated acute myeloid leukemia cells acquired sensitivity to glucocorticoids. Therefore, dexamethasone might sensitize leukemic stem cells to chemotherapy-induced cell death and thus limit the risk of relapse.

This study consists of a screening period, a treatment period, and a post-treatment follow-up period. Adult patients with relapsed/refractory acute myeloid leukemia are randomly assigned in a 1:1 ratio to receive either standard salvage therapy in combination with dexamethasone or standard salvage therapy alone. Standard salvage therapy is intensive chemotherapy (amsacrine-cytarabine) or azacitidine according to the investigator's willingness. For those patients with intensive chemotherapy amsacrine-cytarabine, the study treatment period includes 1 induction cycle and up to 3 consolidation cycles. For those patients with azacitidine, the study treatment period includes 3 cycles prior to the evaluation of the complete remission and thereafter lasts until progression. Of note, any patients in the study can undergo allogeneic hematopoietic stem cell transplantation providing his/her disease is controlled. After discontinuing the study treatment all patients must further carry out post-treatment follow-up visits every 3 months during the first and second year, and every 6 months thereafter until death, withdrawal of consent, loss to follow-up, or the end of the study, whichever occurs first. The end of the study is planned 5 years after the randomization of the first patient. The primary endpoint is the overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age or older
2. Diagnosis of acute myeloid leukemia by World Health Organization classification

   First relapsed or refractory acute myeloid leukemia with at least 5% blasts by bone marrow biopsy or aspirate, or at least 1% blasts in peripheral blood, and meeting the following criteria:

   First relapsed acute myeloid leukemia :
   * First relapse occurred at least 90 days to 24 months after the first complete remission or complete remission with incomplete recovery
   * The first complete remission or complete remission with incomplete recovery had to result from no more than 2 cycles of cytotoxic chemotherapy. At least 1 induction cycle must have consisted of an anthracycline and cytarabine combination with a reasonable schedule/dose of anthracycline in the judgment of the investigator.
   * The re-emergence of at least 5% leukemic blasts in bone marrow is not attributable to other causes, regardless of new or recurrent dysplastic changes or extramedullary disease, or the re-emergence of at least 1% blasts in the peripheral blood is not attributable to other causes such as regenerating marrow.

   Refractory acute myeloid leukemia :
   * Persistent acute myeloid leukemia was documented by bone marrow biopsy or aspirate at least 28 days after day 1 of the first induction cycle of 1 or 2 cycles of cytotoxic chemotherapy.
   * Re-emergence of at least 5% leukemic blasts in bone marrow or at least 1% blasts in peripheral blood is not attributable to other causes such as regenerating marrow, and was less than 90 days after the first complete remission or complete remission with incomplete recovery.
   * Prior induction therapy had to include no more than 2 cycles of cytotoxic chemotherapy. At least 1 induction cycle must have consisted of an anthracycline and cytarabine combination with a reasonable schedule/dose of anthracycline in the judgment of the investigator.
3. Eastern Cooperative Oncology Group performance status ≤ 2.
4. Left ventricular ejection fraction ≥ 50% by echocardiogram or multi-gated acquisition scan ; only applicable for patients who will receive intensive chemotherapy.
5. Serum creatinine ≤ 150 µmol/L and/or total bilirubin ≤ 1.5 × the upper limit of normal and/or, aspartate aminotransferase ≤ 2.5 × the upper limit of normal, and/or alanine aminotransferase ≤ 2.5 × the upper limit of normal (unless related to acute myeloid leukemia)
6. Any clinically significant non-hematological toxicity after prior chemotherapy must be resolved or of grade 1 as per Common Terminology Criteria for Adverse Events version 4.03.
7. Women must be surgically or biologically sterile, or in post-menopause (amenorrheic for at least 12 months), or if of childbearing potential, must have a negative urine or serum pregnancy test within 14 days prior to the randomization and agree to use a highly effective method of contraception throughout the entire duration of the study treatment (including dose interruptions) and until 3 months after the last study treatment administration. Men must be surgically or biologically sterile, or agree to use a highly effective method of contraception throughout the entire duration of the study treatment (including dose interruptions) and until 6 months after the last study treatment administration.
8. Registered to, or beneficiary of, social security insurance or equivalent.
9. Signed written informed consent by both the patient and the investigator prior to perform any study-relayed procedure not part of normal medical care.

Exclusion Criteria:

1. Acute promyelocytic leukemia (M3 subtype of acute myeloid leukemia).
2. More than 2 cycles of first line induction chemotherapy.
3. Acute myeloid leukemia with Philadelphia chromosome or BCR-ABL1 or blast crisis stage of chronic myeloid leukemia.
4. Known or suspected central nervous system leukemia.
5. Undergoing allogeneic hematopoietic stem cell transplantation within 90 days prior to randomization, or being on immunosuppressive therapy for prophylaxis of graft-versus-host disease, or experiencing graft-versus-host disease within 2 weeks prior to randomization.
6. Use of any experimental, cytotoxic, or targeted, anti-leukemic therapy within 14 days prior to randomization, with the exception of hydroxyurea.
7. Formal contraindication to glucocorticoids.
8. Non-acute myeloid leukemia-associated organic or psychiatric severe disease that contraindicates use of study treatment.
9. Patient who may not be followed regularly in consultation because of psychological, family, social, or geographical reasons.
10. History of uncontrolled other malignancy for at least two years, with the exception of basal cell carcinoma and in situ cervix carcinoma.
11. Severe uncontrolled infection at time of inclusion.
12. Positive serology for human immunodeficiency virus-1 or 2, and/or Human T-Cell lymphotropic viruses-1 or 2, and/or active viral infection with hepatitis B virus and/or hepatitis C virus.
13. Pregnant (beta gonadotropic chorionic hormon positive) or breastfeeding woman.
14. Incapable patient of age, under guardianship, under curators or safeguard of justice.
15. Patient under State Medical Assistance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 60 months
  Time from the date of randomization to the date of death from any cause

SECONDARY OUTCOMES:
Response to therapy | Up to 60 months
  Best response of complete remission or complete remission with incomplete recovery as assessed by the investigators according to the 2010 European Leukemia Net recommendations for diagnosis and management of acute myeloid leukemia in adults
Minimal residual disease positivity | Up to 60 months
  Quantitative assessment by either quantitative polymerase chain reaction or multiparameter flow cytometry of any tumor cells greater than pre-specified sensitivity thresholds of detection
Number of patient who realize allogeneic hematopoietic stem cell transplantation | Up to 60 months
  Undergoing allogeneic hematopoietic stem cell transplantation
Duration of remission | Up to 60 months
  Time from the date of first complete remission or complete remission with incomplete recovery to the date of relapse, where complete remission, complete remission with incomplete recovery, and relapse as assessed by the investigators according to the 2010 European Leukemia Net recommendations for diagnosis and management of acute myeloid leukemia in adults
Relapse-free survival | Up to 60 months
  Time from the date of first complete remission or complete remission with incomplete recovery to the date of relapse or death from any cause, whichever occurs first, where complete remission, complete remission with incomplete recovery, and relapse as assessed by the investigators according to the 2010 European Leukemia Net recommendations for diagnosis and management of acute myeloid leukemia in adults
Event-free survival | Up to 60 months
  Time from the date of randomization to the date of treatment failure, or relapse from complete remission or complete remission with incomplete recovery, or death from any cause, whichever occurs first, where treatment failure, complete remission, complete remission with incomplete recovery, and relapse as assessed by the investigators according to the 2010 European Leukemia Net recommendations for diagnosis and management of acute myeloid leukemia in adults
Quality of life with leukemia questionnaire | At baseline, through complete remission, on Day 1 before dosing of each post-remission cycle, at 60 months
  Scoring of functional assessment of cancer therapy - Leukemia questionnaire
Adverse events | During 60 months
  Adverse events reported according to the descriptions and grading scale found in the version 4.03 of the National Cancer Institute - Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Christian RECHER, PhD, Study Director — University Hospital, Toulouse
Locations (10):
- France (10):
  - CH de la Côte Basque, Bayonne, France
  - CHU de la Réunion, Saint-Pierre, France
  - CHU de Grenoble, Grenoble
  - CHU de Limoges, Limoges
  - Institut Paoli Calmettes, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU de Nîmes, Nîmes
  - CHU de Bordeaux, Pessac
  - CHU de Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No